CLINICAL TRIAL: NCT03700580
Title: Application of a Double Blind Clinical Trial Protocol for Evaluation of Healing Action of P1G10, From V Cundinamarcensis to Chronic Neuropathic Wounds in Diabetic Foot Ulcers.
Brief Title: Clinical Trial Using the Proteolytic Fraction P1G10 From V. Cundinamarcensis to Heal Diabetic Foot Ulcer
Acronym: P1G10
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Carlos E Salas (Other)
Responsible Party: Sponsor-Investigator, Carlos E Salas, Professor of Biochemistry, Federal University of Minas Gerais
Organization: Federal University of Minas Gerais (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P1G10
Record Dates: First submitted 2018-10-04; First posted 2018-10-09 (Actual); Last update posted 2018-10-10 (Actual); Status verified 2018-10

CONDITIONS: Diabetic Foot; Neuropathy, Diabetic; Foot Ulcer
Keywords: diabetes type 2; wound healing; peripheral neuropathy; P1G10
MeSH Terms: conditions — Diabetic Foot; Diabetic Neuropathies; Foot Ulcer; Diabetes Mellitus, Type 2; Peripheral Nervous System Diseases

STUDY DESIGN:
Intervention Model Description: The intervention encompassed a topical application on the ulcer bed of the active fraction 0.1% P1G10 dispersed in hydrosoluble vehicle. The control group received hydrogel with the same frequency adopted for P1G10 (Three times per week during 16 weeks). Regardless the intervention prior to each application the ulcer bed was cleaned with 0.9% physiological serum without antiseptic.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hydrogel treatment (Active Comparator): It refers to the standard treatment currently applied for foot ulcers at the Health Center where the study was conducted. The intervention was applied to the cohort, three times a week during 16 weeks or when the wound attained full epithelization. The wound bed was cleaned with physiological serum before application of Hydrogel.
  Interventions: Drug: Hydrogel treatment
- P1G10 treatment (Experimental): It refers to the experimental parallel intervention consisting of three weekly applications of 0.1% P1G10 dispersed in the hydrosoluble vehicle during a 16-week period, or until full epithelization of the wound. The wound bed was cleaned with physiological serum before application of the drug.
  Interventions: Drug: P1G10

INTERVENTIONS:
Drug: Hydrogel treatment — Hydrogel dressing containing water, carboxymethyl cellulose and sodium alginate in non-specified proportions, purchased in bulk amounts was sterile dispensed in smaller amounts (200 g) for frequent use.
  Other Names: Gel Comfeel ®; Coloplast; Hydrogel Purilon ®
  Arms: Hydrogel treatment
Drug: P1G10 — P1G10 containing dressing composed by 8% Polawax, 6% liquid vaseline, 0.06% butylated hydroxytoluene, 0.15% Nipagin, 5% propyleneglycol, 0.1% Nipazol, 0.1% ethylenediaminetetraacetate disodium salt, 0.03% methyl-aminopropanol-95, 0.3% Imidazolidinyl urea, 2% Cyclomethicone, 78.2% distilled water. A single batch of the formulation was made and used throughout the intervention. A sample of this preparation was used to assess the extended stability of the formulation. The formulation was dispensed into 100 g dispensers for weekly use.
  Arms: P1G10 treatment

SUMMARY:
The aim of the study was to investigate the role of the proteolytic fraction from Vasconcellea cundinamarcensis, designated as P1G10, on healing of chronic foot ulcers in neuropathic patients diagnosed with diabetes type 2. Fifty patients were enrolled in a prospective, randomized, double-blind trial, to verify the efﬁcacy and safety of a topical dressing containing 0.1% P1G10, versus a Hydrogel (positive control) protocol currently applied at the Health Center to treat this condition. Upon completion of the intervention, the outcome evaluated the number of patients attaining full epithelization (100%), or at least 80% healing in both arms (P1G10 versus Hydrogel). Statistical analysis compared the endpoint data on each group to assess the signiﬁcance of differences.

DETAILED DESCRIPTION:
Volunteers admitted for the study were randomly assigned into two distinct treatment groups. Randomization was performed by simple and stratified draw for each type of treatment. The treatment options were: a) Hydrogel™ and b) P1G10. The active principle had been previously dissolved in water and dispersed into Polawax dressing at 0.1% w/w final. Polawax™ is an emulsifying wax for cosmetic preparations. According to the manufacturers, it is able to hold together all types of ingredients without residue or separation. It is, therefore, ideal for "oil in water" creams and lotions. Number were used to identify both formulations.

The staff participating in this clinical trial, including researchers was unaware of the identity of the formulation applied on each proband. Each formulation used during the intervention was dispensed weekly at the Laboratory of Antitumor Substances of the Institute of Biological Sciences of the Federal University of Minas Gerais by members of the research group who had no contact with the staff responsible for the application of the protocol. The formulations were stored at 4°C until its application.

The treatment and the collection of data, took place between August 2012 and October 2016, and it was carried out by health professional and a technical assistant previously trained to evaluate and perform the procedure.

The application of the intervention was done three times per week (Monday, Wednesday and Friday), completing 48 applications or until full epithelialization of the ulcer was observed, whichever occurred first. The treatment was performed exclusively at the outpatient level. When the proband could not attend the scheduled treatment, he (she) was instructed to perform the dressing change only with 0.9% saline solution. Patients who missed two consecutive scheduled interventions were withdrawn from the study.

Ulcers were cleaned with 0.9% physiological solution using soft pressure, without scrubbing or addition of antiseptic substances. Subsequently, a thin layer of the ointment containing P1G10 or Hydrogel was applied over the ulcer bed, covering all its extension. Then double gauze was applied, fixed with adhesive tape and crepe bandage, if necessary. In cases of users with more than one wound, each wound received identical treatment, but only one ulcer was selected for the study.

During the first week of treatment, the subjects were observed for 30 minutes after the intervention, in order to verify possible undesirable effects. After this interval, if they did not present adverse events, they were released. Users were also instructed to contact the responsible investigators by telephone if they observed the emergence of any adverse effects. A prior trial of the formulation containing 0.1% P1G10 applied onto the arm of healthy individuals during one-month did not induce local or systemic affects.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of diabetes 2 had
* Hemoglobin ≥ 9.0 g/dl
* total leukocytes ≥ 300/ mm3
* platelets ≥ 100.00/mm3
* total bilirubin ≤ 1.0 mg/dL
* aspartate aminotransferase between 14 and 17 U/L in males and 10 and 33 U/L in females
* pyruvate transaminase between 10 and 40 U/L in males and 7 and 35 U/L in females
* creatinine between 0.70 and 1.20 mg/dL in males and 0.6 and 1.0 mg/dL in females

Exclusion criteria

* pregnant females
* lactating mothers
* highly exuding ulcers
* patients receiving alternative treatments for ulcers
* reported allergy to the components included in the formulation,
* concomitant uncontrolled morbidity
* current active infections,
* HIV serum positives
* diagnosed with neoplasia or undergoing treatment with a cytostatic, or immunosuppressing agent
* individuals subjected to radiotherapy within the last 3 months before beginning the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2012-08-15 (Actual); Primary Completion 2016-10-14 (Actual); Study Completion 2016-10-15 (Actual)

PRIMARY OUTCOMES:
100% epithelization | The primary outcome (100% epithelization) is measured at the time of the intervention (1-16 weeks). If this endpoint is attained at a given date, the interval between the first intervention and the endpoint date is the period scored for the event.
  A primary end point was considered as full re-epithelization (100%) of the injury assessed by presence of epithelial tissue in 100% of the bed occurring during, or at the end of 48 applications. Quantification of healing is assessed by measure of the wound area, registered with Sony camera (Cyber-shot), 18.2 megapixels. Along the ulcer is positioned a standard mold (5.1 x 15.0) cm including proband's initials, record number and date of treatment. A transparent sterile paper superimposed on the wound, measured the orthogonal lengths to estimate the wound area. Normal distribution of data was evaluated with Shapiro-Wilk test. The differences in values between groups were assessed by t- test. Wound healing incidence was expressed as 1000 person-day with 95% confidence interval in both groups. To minimize the effect of noncompliance and missing outcomes, the data were analyzed as "intention to treat" thus including every subject enrolled in each group during the initial assignment.

SECONDARY OUTCOMES:
80% epithelization | The secondary outcome (80% epithelization) is measured at the time of the intervention (1-16 weeks). If this endpoint is attained at a given date, the interval between the first intervention and the endpoint date is the period scored for the event.
  A secondary end point was considered as 80% re-epithelization of the injury assessed by presence of epithelial tissue in 80% of the bed occurring during, or at the end of 48 applications. Quantification of healing is assessed by measure of the wound area, registered with Sony camera (Cyber-shot), 18.2 megapixels. Along the ulcer is positioned a standard mold (5.1 x 15.0) cm including proband's initials, record number and date of treatment. A transparent sterile paper superimposed on the wound measured the orthogonal lengths to estimate the wound area. Normal distribution of data was evaluated with Shapiro-Wilk test. The differences in values between groups were assessed by t- test. Wound healing incidence was expressed as 1000 person-day with 95% confidence interval in both groups. To minimize the effect of noncompliance and missing outcomes, the data were analyzed as "intention to treat" thus including every subject enrolled in each group during the initial assignment.

CONTACTS AND LOCATIONS:
Overall Officials: Miriam T Lopes, PhD, Study Director — Federal University of Minas Gerais
Locations (1):
- Unidade de Referência Secundária (URS) Padre Eustáquio, do Distrito Sanitário Noroeste da Secretaria Municipal e Saúde de Belo Horizonte., Belo Horizonte, Minas Gerais, Brazil

REFERENCES:
- [Background] Freitas KM, Barcelos LS, Caliari MV, Salas CE, Lopes MTP. Healing activity of proteolytic fraction (P1G10) from Vasconcellea cundinamarcensis in a cutaneous wound excision model. Biomed Pharmacother. 2017 Dec;96:269-278. doi: 10.1016/j.biopha.2017.09.109. Epub 2017 Oct 6. PMID 28988012
- [Result] Tonaco LAB, Gomes FL, Velasquez-Melendez G, Lopes MTP, Salas CE. The Proteolytic Fraction from Latex of Vasconcellea cundinamarcensis (P1G10) Enhances Wound Healing of Diabetic Foot Ulcers: A Double-Blind Randomized Pilot Study. Adv Ther. 2018 Apr;35(4):494-502. doi: 10.1007/s12325-018-0684-2. Epub 2018 Mar 21. PMID 29564750